CLINICAL TRIAL: NCT05264220
Title: Exploring the Effects of a Brief Values-Based Intervention on Adherence to Fluid Restriction Recommendations and Quality of Life in Haemodialysis Patients
Brief Title: Fluid Restriction and Quality of Life on Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); Oxford Health NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PID15290
Record Dates: First submitted 2022-01-13; First posted 2022-03-03 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-01

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Single group study - multiple baseline case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT Matrix (Experimental): Participants will each receive the ACT Matrix intervention. Participants will be randomised to multiple start dates, producing different baseline durations.
  Interventions: Behavioral: ACT Matrix

INTERVENTIONS:
Behavioral: ACT Matrix — Participants will receive a 4 session psychological intervention based on the ACT Matrix

SUMMARY:
Almost 30,000 people in the UK receive dialysis due to end stage renal disease (ESRD). Although dialysis prolongs life, people receiving dialysis are still typically bothered by a range of physical symptoms and need to make substantial adjustments in order to accommodate ESRD and its treatment. One adjustment that is often required is a dramatic reduction in fluid intake. Although sticking to fluid intake restrictions improves the efficiency of dialysis, monitoring fluid intake is complicated. The restrictions also leave people feeling very thirsty so restrictions can be hard to stick to. This project will develop and test a brief psychological intervention for people who struggle to adhere to fluid intake restrictions and will aim to increase quality of life whilst on dialysis. The intervention will be developed with input from people with lived experience of ESRD. It will then be offered to 12 people, recruited from clinics, who will complete questionnaires to monitor experiences and symptoms before, during and after the intervention. Participants' data will be analysed to find out whether the intervention has been helpful in reducing fluid intake and improving quality of life. If the findings are promising, this would suggest that the intervention could be tested in a larger clinical study in the future.

DETAILED DESCRIPTION:
Please note: this study adopts a between-subjects concurrent multiple baseline single case ABC experimental design. Participant change within and across phases A (baseline, variable with participants randomised to a 6, 8, or 10 week baseline), B (4 week intervention phase) and C (4 week follow-up) will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving haemodialysis for end-stage kidney disease
* Aged 18+
* Adequate fluency in written and spoken English to undertake the intervention and complete measures (assessed by research psychologist during discussion of study commitment)
* Willing and able to participate in face-to-face and/or digital delivery of a psychological intervention (e.g. if digital delivery is requested or/or necessitated by Covid 19 restrictions patient has access to a computer, tablet or phone).
* Identified by clinical staff as having difficulty with adherence to fluid intake recommendations.
* Consents to participation, including recording of video sessions for fidelity/adherence rating and supervision.

Exclusion Criteria:

* • Lack of capacity to consent

  * Poorly controlled diabetes resulting in recent hospital admissions for hypo/hyperglycaemic episode(s)
  * Intellectual disability that prevents self-management of fluid intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Dialysis Diet and Fluid Intake Non-Adherence Questionnaire (Vlamink et al., 2001) | baseline phase week 2
  This brief four-item measure assesses adherence to diet and fluid requirements over the previous 14 days. It includes the following items: 1) On how many days during the last 14 didn't you follow your diet guidelines? 2) To what degree did you deviate from your diet guidelines? (0-no deviation to 4 - very severe deviation) 3) On how many days during the last 14 didn't you follow your fluid guidelines? 4) To what degree did you deviate from your fluid guidelines? (0-no deviation to 4 - very severe deviation).
Dialysis Diet and Fluid Intake Non-Adherence Questionnaire (Vlamink et al., 2001) | baseline phase week 4
  This brief four-item measure assesses adherence to diet and fluid requirements over the previous 14 days. It includes the following items: 1) On how many days during the last 14 didn't you follow your diet guidelines? 2) To what degree did you deviate from your diet guidelines? (0-no deviation to 4 - very severe deviation) 3) On how many days during the last 14 didn't you follow your fluid guidelines? 4) To what degree did you deviate from your fluid guidelines? (0-no deviation to 4 - very severe deviation).
Dialysis Diet and Fluid Intake Non-Adherence Questionnaire (Vlamink et al., 2001) | baseline phase week 6
  This brief four-item measure assesses adherence to diet and fluid requirements over the previous 14 days. It includes the following items: 1) On how many days during the last 14 didn't you follow your diet guidelines? 2) To what degree did you deviate from your diet guidelines? (0-no deviation to 4 - very severe deviation) 3) On how many days during the last 14 didn't you follow your fluid guidelines? 4) To what degree did you deviate from your fluid guidelines? (0-no deviation to 4 - very severe deviation).
Dialysis Diet and Fluid Intake Non-Adherence Questionnaire (Vlamink et al., 2001) | baseline phase week 8 (those randomised to 8 and 10 week baselines only)
  This brief four-item measure assesses adherence to diet and fluid requirements over the previous 14 days. It includes the following items: 1) On how many days during the last 14 didn't you follow your diet guidelines? 2) To what degree did you deviate from your diet guidelines? (0-no deviation to 4 - very severe deviation) 3) On how many days during the last 14 didn't you follow your fluid guidelines? 4) To what degree did you deviate from your fluid guidelines? (0-no deviation to 4 - very severe deviation).
Dialysis Diet and Fluid Intake Non-Adherence Questionnaire (Vlamink et al., 2001) | baseline phase week 10 (those randomised to 10 week baseline only)
  This brief four-item measure assesses adherence to diet and fluid requirements over the previous 14 days. It includes the following items: 1) On how many days during the last 14 didn't you follow your diet guidelines? 2) To what degree did you deviate from your diet guidelines? (0-no deviation to 4 - very severe deviation) 3) On how many days during the last 14 didn't you follow your fluid guidelines? 4) To what degree did you deviate from your fluid guidelines? (0-no deviation to 4 - very severe deviation).
Dialysis Diet and Fluid Intake Non-Adherence Questionnaire (Vlamink et al., 2001) | intervention phase week 2
  This brief four-item measure assesses adherence to diet and fluid requirements over the previous 14 days. It includes the following items: 1) On how many days during the last 14 didn't you follow your diet guidelines? 2) To what degree did you deviate from your diet guidelines? (0-no deviation to 4 - very severe deviation) 3) On how many days during the last 14 didn't you follow your fluid guidelines? 4) To what degree did you deviate from your fluid guidelines? (0-no deviation to 4 - very severe deviation).
Dialysis Diet and Fluid Intake Non-Adherence Questionnaire (Vlamink et al., 2001) | intervention phase week 4
  This brief four-item measure assesses adherence to diet and fluid requirements over the previous 14 days. It includes the following items: 1) On how many days during the last 14 didn't you follow your diet guidelines? 2) To what degree did you deviate from your diet guidelines? (0-no deviation to 4 - very severe deviation) 3) On how many days during the last 14 didn't you follow your fluid guidelines? 4) To what degree did you deviate from your fluid guidelines? (0-no deviation to 4 - very severe deviation).
Dialysis Diet and Fluid Intake Non-Adherence Questionnaire (Vlamink et al., 2001) | 4 week (from end of intervention) follow-up
  This brief four-item measure assesses adherence to diet and fluid requirements over the previous 14 days. It includes the following items: 1) On how many days during the last 14 didn't you follow your diet guidelines? 2) To what degree did you deviate from your diet guidelines? (0-no deviation to 4 - very severe deviation) 3) On how many days during the last 14 didn't you follow your fluid guidelines? 4) To what degree did you deviate from your fluid guidelines? (0-no deviation to 4 - very severe deviation).
Interdialytic weight gain | Baseline phase week 1
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.
Interdialytic weight gain | Baseline phase week 2
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.
Interdialytic weight gain | Baseline phase week 3
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.
Interdialytic weight gain | Baseline phase week 4
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.
Interdialytic weight gain | Baseline phase week 5
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.
Interdialytic weight gain | Baseline phase week 6
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.
Interdialytic weight gain | Baseline phase week 7 (those randomised to 8 or 10 week follow-up)
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.
Interdialytic weight gain | Baseline phase week 8 (those randomised to 8 or 10 week follow-up)
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.
Interdialytic weight gain | Baseline phase week 9 (those randomised to 10 week baselines)
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.
Interdialytic weight gain | Baseline phase week 10 (those randomised to 10 week baseline)
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.
Interdialytic weight gain | intervention week 1
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.
Interdialytic weight gain | intervention week 2
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.
Interdialytic weight gain | intervention week 3
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.
Interdialytic weight gain | intervention week 4
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.
Interdialytic weight gain | four week follow-up
  participant's interdialytic weight gain between each dialysis session will be obtained from medical records if possible.

SECONDARY OUTCOMES:
Valuing Questionnaire | baseline week 1
  This 10-item questionnaire assesses wellbeing as it relates to a person's ability to live the kind of life they value. It is designed for weekly administration. Items include statements such as "I made progress in the areas of life I care most about" and "my behaviour was a good example of what I stand for in life". Each item is rated on a scale ranging from 1 (not at all true) to 7 (completely true).
Valuing Questionnaire | baseline week 2
  This 10-item questionnaire assesses wellbeing as it relates to a person's ability to live the kind of life they value. It is designed for weekly administration. Items include statements such as "I made progress in the areas of life I care most about" and "my behaviour was a good example of what I stand for in life". Each item is rated on a scale ranging from 1 (not at all true) to 7 (completely true).
Valuing Questionnaire | baseline week 3
  This 10-item questionnaire assesses wellbeing as it relates to a person's ability to live the kind of life they value. It is designed for weekly administration. Items include statements such as "I made progress in the areas of life I care most about" and "my behaviour was a good example of what I stand for in life". Each item is rated on a scale ranging from 1 (not at all true) to 7 (completely true).
Valuing Questionnaire | baseline week 4
  This 10-item questionnaire assesses wellbeing as it relates to a person's ability to live the kind of life they value. It is designed for weekly administration. Items include statements such as "I made progress in the areas of life I care most about" and "my behaviour was a good example of what I stand for in life". Each item is rated on a scale ranging from 1 (not at all true) to 7 (completely true).
Valuing Questionnaire | baseline week 5
  This 10-item questionnaire assesses wellbeing as it relates to a person's ability to live the kind of life they value. It is designed for weekly administration. Items include statements such as "I made progress in the areas of life I care most about" and "my behaviour was a good example of what I stand for in life". Each item is rated on a scale ranging from 1 (not at all true) to 7 (completely true).
Valuing Questionnaire | baseline week 6
  This 10-item questionnaire assesses wellbeing as it relates to a person's ability to live the kind of life they value. It is designed for weekly administration. Items include statements such as "I made progress in the areas of life I care most about" and "my behaviour was a good example of what I stand for in life". Each item is rated on a scale ranging from 1 (not at all true) to 7 (completely true).
Valuing Questionnaire | baseline week 7 (those randomised to 8 and 10 week baselines only)
  This 10-item questionnaire assesses wellbeing as it relates to a person's ability to live the kind of life they value. It is designed for weekly administration. Items include statements such as "I made progress in the areas of life I care most about" and "my behaviour was a good example of what I stand for in life". Each item is rated on a scale ranging from 1 (not at all true) to 7 (completely true).
Valuing Questionnaire | baseline week 8 (those randomised to 8 and 10 week baselines only)
  This 10-item questionnaire assesses wellbeing as it relates to a person's ability to live the kind of life they value. It is designed for weekly administration. Items include statements such as "I made progress in the areas of life I care most about" and "my behaviour was a good example of what I stand for in life". Each item is rated on a scale ranging from 1 (not at all true) to 7 (completely true).
Valuing Questionnaire | baseline week 9 (those randomised to 10 week baselines only)
  This 10-item questionnaire assesses wellbeing as it relates to a person's ability to live the kind of life they value. It is designed for weekly administration. Items include statements such as "I made progress in the areas of life I care most about" and "my behaviour was a good example of what I stand for in life". Each item is rated on a scale ranging from 1 (not at all true) to 7 (completely true).
Valuing Questionnaire | baseline week 10 (those randomised to 10 week baselines only)
  This 10-item questionnaire assesses wellbeing as it relates to a person's ability to live the kind of life they value. It is designed for weekly administration. Items include statements such as "I made progress in the areas of life I care most about" and "my behaviour was a good example of what I stand for in life". Each item is rated on a scale ranging from 1 (not at all true) to 7 (completely true).

OTHER OUTCOMES:
End-Stage Renal Disease Adherence Questionnaire (ESRD-AQ; Kim et al., 2010) | Study intake assessment
  This self-report measure includes 46 questions assessing adherence to medication, diet, fluid intake restrictions and participation in dialysis sessions. It has excellent psychometric properties.
The Clinical Outcomes Routine Evaluation (CORE) -10 (Barkham et al., 2013) | Baseline week 1
  This measure assesses severity of clinical symptoms, across 10 items, each rated 0-4. The measure differentiates clinical samples from non-clinical populations. It has adequate convergent validity when correlated with other clinical measures, and good internal reliability (Cronbach's alpha > .80) and sensitivity to change (see Connell & Barkham, 2007). A change on the CORE-10 of six or more points corresponds to statistically reliable change. Scores on the measure are interpreted as follows: 0-5 (healthy); 6-10 (low level); 11-15 (mild); 16-20 (moderate); 21-25 (moderately severe); 26 + (severe).
The Clinical Outcomes Routine Evaluation (CORE) -10 (Barkham et al., 2013) | intervention week 1
  This measure assesses severity of clinical symptoms, across 10 items, each rated 0-4. The measure differentiates clinical samples from non-clinical populations. It has adequate convergent validity when correlated with other clinical measures, and good internal reliability (Cronbach's alpha > .80) and sensitivity to change (see Connell & Barkham, 2007). A change on the CORE-10 of six or more points corresponds to statistically reliable change. Scores on the measure are interpreted as follows: 0-5 (healthy); 6-10 (low level); 11-15 (mild); 16-20 (moderate); 21-25 (moderately severe); 26 + (severe).
The Clinical Outcomes Routine Evaluation (CORE) -10 (Barkham et al., 2013) | intervention week 4
  This measure assesses severity of clinical symptoms, across 10 items, each rated 0-4. The measure differentiates clinical samples from non-clinical populations. It has adequate convergent validity when correlated with other clinical measures, and good internal reliability (Cronbach's alpha > .80) and sensitivity to change (see Connell & Barkham, 2007). A change on the CORE-10 of six or more points corresponds to statistically reliable change. Scores on the measure are interpreted as follows: 0-5 (healthy); 6-10 (low level); 11-15 (mild); 16-20 (moderate); 21-25 (moderately severe); 26 + (severe).
The Clinical Outcomes Routine Evaluation (CORE) -10 (Barkham et al., 2013) | Four week follow-up
  This measure assesses severity of clinical symptoms, across 10 items, each rated 0-4. The measure differentiates clinical samples from non-clinical populations. It has adequate convergent validity when correlated with other clinical measures, and good internal reliability (Cronbach's alpha > .80) and sensitivity to change (see Connell & Barkham, 2007). A change on the CORE-10 of six or more points corresponds to statistically reliable change. Scores on the measure are interpreted as follows: 0-5 (healthy); 6-10 (low level); 11-15 (mild); 16-20 (moderate); 21-25 (moderately severe); 26 + (severe).
EQ-5D-5L (EuroQuol Group, 2009). | Baseline phase week 1
  This widely used measure assesses quality of life across five domains: mobility, self-care, usual activities, pain / discomfort, anxiety/depression. Each domain is rated on a five-level scale: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. Additionally, respondents complete a health thermometer rating their current health status on a scale from 0 to 100. The EQ-5D-5L is a widely used measure for assessing health status with normative data available for UK samples.
EQ-5D-5L (EuroQuol Group, 2009). | Intervention week 1
  This widely used measure assesses quality of life across five domains: mobility, self-care, usual activities, pain / discomfort, anxiety/depression. Each domain is rated on a five-level scale: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. Additionally, respondents complete a health thermometer rating their current health status on a scale from 0 to 100. The EQ-5D-5L is a widely used measure for assessing health status with normative data available for UK samples.
EQ-5D-5L (EuroQuol Group, 2009). | Intervention week 4
  This widely used measure assesses quality of life across five domains: mobility, self-care, usual activities, pain / discomfort, anxiety/depression. Each domain is rated on a five-level scale: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. Additionally, respondents complete a health thermometer rating their current health status on a scale from 0 to 100. The EQ-5D-5L is a widely used measure for assessing health status with normative data available for UK samples.
EQ-5D-5L (EuroQuol Group, 2009). | Four week follow-up
  This widely used measure assesses quality of life across five domains: mobility, self-care, usual activities, pain / discomfort, anxiety/depression. Each domain is rated on a five-level scale: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. Additionally, respondents complete a health thermometer rating their current health status on a scale from 0 to 100. The EQ-5D-5L is a widely used measure for assessing health status with normative data available for UK samples.
Dialysis Symptoms Index (Weisbord et al., 2004) | Baseline week 1
  Measure of common physical and psychological symptoms experienced by people on dialysis
Dialysis Symptoms Index (Weisbord et al., 2004) | Intervention week 1
  Measure of common physical and psychological symptoms experienced by people on dialysis
Dialysis Symptoms Index (Weisbord et al., 2004) | Intervention week 4
  Measure of common physical and psychological symptoms experienced by people on dialysis
Dialysis Symptoms Index (Weisbord et al., 2004) | Four week follow-up
  Measure of common physical and psychological symptoms experienced by people on dialysis
CompACT (Francis, Dawson & Golijani-Moghaddam, 2016) | Baseline week 1
  This 23-item questionnaire assesses psychological flexibility. In addition to a total score, three subscale scores reflecting openness to experience, behavioural awareness and valued action can be derived. Each item is rated on a scale ranging from 0 (strongly disagree) to 6 (strongly agree).
CompACT (Francis, Dawson & Golijani-Moghaddam, 2016) | Intervention week 1
  This 23-item questionnaire assesses psychological flexibility. In addition to a total score, three subscale scores reflecting openness to experience, behavioural awareness and valued action can be derived. Each item is rated on a scale ranging from 0 (strongly disagree) to 6 (strongly agree).
CompACT (Francis, Dawson & Golijani-Moghaddam, 2016) | Intervention week 4
  This 23-item questionnaire assesses psychological flexibility. In addition to a total score, three subscale scores reflecting openness to experience, behavioural awareness and valued action can be derived. Each item is rated on a scale ranging from 0 (strongly disagree) to 6 (strongly agree).
CompACT (Francis, Dawson & Golijani-Moghaddam, 2016) | Four week follow-up
  This 23-item questionnaire assesses psychological flexibility. In addition to a total score, three subscale scores reflecting openness to experience, behavioural awareness and valued action can be derived. Each item is rated on a scale ranging from 0 (strongly disagree) to 6 (strongly agree).
Intervention Credibility/Expectancy Questionnaire (Devilly & Borkovec, 2000) | Intervention week 1
  measure of participants' views on intervention credibility
Intervention Credibility/Expectancy Questionnaire (Devilly & Borkovec, 2000) | Four week follow-up
  measure of participants' views on intervention credibility

CONTACTS AND LOCATIONS:
Overall Officials: Catherine H Crane, DPhil, Principal Investigator — University of Oxford
Locations (1):
- Renal and Transplant Medicine Unit (and satellite units), Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom